CLINICAL TRIAL: NCT07035028
Title: Evaluation of Fetal Response to Intrapartum Digital Fetal Scalp Stimulation Upon Detection of Suspected Loss of Fetal Well-being in Suspicious and Pathologic Cardiotocographic Recordings, to Identify Intrapartum Fetal Hypoxia.
Brief Title: Evaluation of the Fetal Response to Intrapartum Digital Fetal Scalp Stimulation to Identify Intrapartum Fetal Hypoxia.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: CEU San Pablo University (Other); Hospital Universitario Sanitas La Zarzuela (Other)
Responsible Party: Principal Investigator, Raquel Maqueda Moreno, Investigator name, Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PIC005-24_FJD
Record Dates: First submitted 2025-05-29; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Fetal Hypoxia; Fetal Monitoring
Keywords: digital fetal scalp stimulation dFSS; fetal monitoring; fetal blood sampling FBS; fetal scalp blood; cardiotocography; umbilical cord blood; acidemia; Intrapartum care
MeSH Terms: conditions — Fetal Hypoxia

STUDY DESIGN:
Intervention Model Description: Control group Experimental group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- digital fetal scalp stimulation dFSS (Experimental): Digital fetal scalp stimulation will be performed for a period of 30 seconds prior to obtaining the fetal blood sample. Digital fetal scalp stimulation will be performed by vaginal touch with a gauze pad and applying rubbing pressure over the fetal scalp for 30 to 60 seconds. This procedure will be recorded on the same RCTG. The FHR pattern on the cardiotocographic recording is closely monitored for 1 to 10 minutes, using a 5-minute mean, following fetal stimulation the fetus should respond with an acceleration of FHR defined as an increase in FHR ≥ 15 bpm (beats per minute for at least 15 seconds or normal FHR variability (5 to 25 bpm), or both. The presence of an acceleration of FHR or an increase in variability when it was previously reduced, or both, is interpreted as a positive response, comparable to a normal fetal blood scalp sample FBS result.
  Interventions: Diagnostic Test: Digital fetal scalp stimulation dFSS
- NO digital fetal scalp stimulation dFSS (No Intervention): The fetal blood sampling will be performed, since in our environment it is the gold standard method included in the SEGO recommendations.
  There is NO intervention.

INTERVENTIONS:
Diagnostic Test: Digital fetal scalp stimulation dFSS — Digital fetal scalp stimulation will be performed for a period of 30 seconds, prior to obtaining the fetal blood sample. Digital fetal scalp stimulation will be performed by vaginal touch with a gauze pad and rubbing the fetal scalp with pressure for 30 to 60 seconds.
  Other Names: dFSS
  Arms: digital fetal scalp stimulation dFSS

SUMMARY:
The main objective of this study is to evaluate whether digital fetal scalp stimulation improves fetal well-being in fetuses with suspicious or pathological cardiotocographic recordings, showing an improvement in cardiotocographic recording patterns and normal values in intrapartum fetal scalp blood results.

Upon detection of a suspicious or pathologic cardiotocographic recording, the investigators need to perform an objective verification of fetal well-being.

Currently, fetal scalp blood is the reference test to assess intrapartum fetal hypoxia, according to the protocols of the Spanish Society of Gynecology and Obstetrics.

This procedure lasts about 5 minutes and consists of taking a small sample of the fetal scalp, through a vaginal exploration, the blood is collected in a thin tube and analyzed by a machine in the delivery room obtaining the results in a few minutes.

The investigators emphasize that this test is not part of the study, as long as the monitor is suspicious or pathological, it will be performed according to protocol to objectively assess fetal well-being.

Currently there are studies that support the use of fetal scalp stimulation as an alternative technique to assess intrapartum fetal well-being and predict neonatal outcomes, but they also highlight its limited evidence.

Digital fetal scalp stimulation is a NON-invasive method, as no instrument is required and fetal stimulation is a 30-60 second surface rubbing pressure, which is performed manually, through vaginal exploration, the same technique the investigators use to assess dilation during the labor process.

Each patient will be randomly assigned to a study group:

Experimental group: before the extraction of capillary blood from the fetal scalp, fetal head stimulation will be performed, a technique that poses no risk to the baby. The researchers need the consent of the participants to perform this technique and collect data.

Control group: fetal head stimulation will not be applied, but data from the clinical history necessary for this study will be collected.

In no case will extraordinary or unnecessary tests be performed for participation in this study.

This study will have an Informed Consent document.

This study will be carried out at the Fundación Jiménez Díaz and Zarzuela and will include 182 patients for 24 months.

DETAILED DESCRIPTION:
The goal of intrapartum care is to ensure excellent maternal and perinatal outcomes. Normal labor is characterized by regular uterine contractions, which cause repeated transient interruptions in fetal oxygenation. Most fetuses tolerate this process well, but some do not. The fetal heart rate (FHR) pattern helps distinguish the former from the latter, as it is an indirect marker of fetal cardiac and central nervous system responses to changes in blood pressure, blood gases, and acid-base status. The term "suspected fetal compromise or risk of loss of fetal well-being" is used in obstetrics, when the fetus is considered to be at increased risk of ischemic hypoxic injury, brain damage or death, and is one of the most common indications for emergency cesarean section during labor. In our setting, continuous electronic fetal heart rate monitoring recorded by cardiotocography (CTG) is routinely used in labor to identify fetuses that may be at increased risk of compromise and may benefit from further evaluation of fetal well-being or other interventions. CTG tracings display the fetal heart rate (FHR) pattern along with maternal uterine activity.

CTG patterns are classified into discrete general categories according to four criteria: basal FHR, heart rate variability, presence or absence of FHR accelerations, and decelerations. An example of such a classification system is the 2015 FIGO International Federation of Gynecology and Obstetrics guideline, on which the investigators will base our study. The Spanish Society of Gynecology and Obstetrics defines the registry in normal, suspicious, and pathologic categories. Regardless of the classification system used, abnormal FHR patterns that do not respond to basic intrauterine resuscitation measures require further evaluation of fetal well-being and/or termination of pregnancy, either by cesarean section, assisted vaginal delivery, or spontaneous vaginal delivery.

CTG has a high false-positive rate for fetal compromise (60%) and the studies of Chandraharan et al are gaining momentum, where intrapartum interventions should be based on a thorough understanding of the features observed on the tracing recordings to differentiate normal fetal response to continued stress from the onset of compensation, so that timely action can be taken to avoid hypoxic ischemic encephalopathy and prenatal deaths, while avoiding unnecessary intrapartum interventions to the mother. Cesarean section rates are increasing worldwide, much of that increase is due to primary cesarean sections among nulliparous women due to emergency procedures in labor. Our great challenge is to achieve a reliable test of fetal well-being during labor and to be able to be minimally invasive for both mother and fetus.

When a suspicious or pathologic FHR pattern is detected and immediate delivery is not warranted, further evaluation of fetal well-being is necessary; such second-line evaluations or tests include fetal scalp blood, in Spain Gold standard to identify fetuses with acidosis and reduce the false positive rate of CTG, and digital fetal scalp stimulation. Clinical guidelines support the use of digital fetal scalp stimulation but also note that research evidence is limited. Digital fetal scalp stimulation is the least invasive method, as it does not require instruments; it involves rubbing the surface of the fetal scalp with pressure for 30 to 60 seconds; the response to stimulation should be evident in cardiotocographic patterns over the next 10 minutes, using a 5-minute average. Fetal scalp stimulation should elicit an acceleration of FHR defined as an increase in FHR ≥ 15 bpm for at least 15 seconds or normal FHR variability (5 to 25 bpm), or both. The presence of an acceleration of FHR or an increase in variability (when previously reduced), or both, is interpreted as a positive response, comparable to a normal fetal scalp blood pH result greater than 7.20.

Fetal scalp blood sampling is an intrapartum procedure to assess the presence and degree of fetal acidemia by analyzing fetal capillary blood for pH or lactate, as both give similar results, with pH being the gold standard test for fetal acidosis in our setting. An amnioscope with a light source is used to expose the fetal scalp, which is cleaned with a 2% aqueous chlorhexidine gauze from blood, mucosa and amniotic fluid, then the scalp is punctured with a 2 mm blade. The blood is collected in long capillary tubes. The test requires the cervix to be dilated at least 2 to 3 cm, can be difficult to perform and may be uncomfortable for the laboring woman. It is contraindicated when the mother is known to have a serious transmissible infection, such as HIV or hepatitis, and in fetuses at increased risk of hemorrhage. Rare complications described in case reports include infection, hemorrhage and cerebrospinal fluid leakage. The procedure will result in stimulation of the fetus, but the primary intent is to collect a scalp blood that will allow quantitative analysis of fetal pH or lactate, reflecting fetal blood oxygenation.

It is not taken into account that the scalp skin is a nonessential peripheral tissue that undergoes catecholamine-induced vasoconstriction early in the fetal stress response and therefore fetal scalp blood sampling does not reflect oxygenation of the fetal central organs and alkaline amniotic fluid and bile acids from meconium may alter results. It has also been shown that fetal scalp blood has no significant effect on the cesarean section rate in women monitored by continuous cardiotocography. Intrapartum fetal scalp blood sampling to measure pH, base excess or deficit, or lactate has not been clearly demonstrated to reduce emergency cesarean deliveries or operative vaginal deliveries or to improve long-term perinatal outcome.

For this reason and many others, such as quality control problems, cost, patient discomfort, sample failure rates of up to 10% and the lack of availability of sampling kits, fetal scalp blood sampling is only rarely performed in the United States and other countries, which is not currently the situation in Spain, since for the SEGO it continues to be the gold standard for detecting fetal acidosis.

The NICE 2022 guideline conducted a review comparing fetal blood sampling with digital fetal scalp stimulation and noted that the studies conducted to date were of low to very low quality, similar to the Cochrane 2023 review which includes two studies Hughes 2022 and Tahmina 2022 , in which Hughes compares fetal scalp stimulation and cardiotocographic patterns with fetal scalp blood samples and cardiotocographic patterns and Tahmina compares fetal head stimulation and cardiotocographic patterns with no fetal head stimulation intervention. The Hughes study reported an apgar score of less than 7 at 5 minutes, a finding that was not recorded in Tahmina, which reported a lower risk of cesarean section in the fetal scalp stimulation group, but again both studies are of very low quality. Although not included in the NICE or Cochrane review, there are other studies that demonstrate that the effectiveness of fetal scalp stimulation is poor for ruling out or confirming fetal hypoxia during labor.

Therefore, very low certainty evidence is available that makes it unclear whether fetal scalp stimulation is a safe and effective way to confirm fetal well-being during labor. Current studies have limitations. More high quality studies with sufficient sample size are needed to evaluate this research question. There is an ongoing study (FIRSST) that will be added to the NICE review in a later update.

The current project aims to give value to a second tier test with little demonstrated scientific evidence, fetal scalp stimulation.

ELIGIBILITY:
Inclusion criteria:

Women with singleton pregnancy.

Cephalic presentation.

Gestational age greater than or equal to 37 weeks.

Pathological cardiotocographic record according to the criteria published by FIGO and with indication to perform a second-line complementary test, in our case a gold standard test of fetal scalp blood FBS, which confirms or not if there is a risk of loss of fetal well-being and the need for fetal extraction.

Signature of HIP and CI for data collection.

Exclusion criteria:

Under 18 years of age.

Contraindication for FBS

Uterine dilatation that does not make FBS possible.

HIV

Hepatitis

Fetuses at increased risk of hemorrhage.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 182 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of fetuses with positive response to digital fetal scalp stimulation, intrapartum ph greater than 7.20, newborn ph greater than 7.20 and good neonatal outcomes | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation, obtain an intrapartum pH greater than 7.20, at birth a pH greater than 7.20, and good neonatal outcomes.

SECONDARY OUTCOMES:
Differences in the cardiotocographic pattern of fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in the cardiotocographic pattern of fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation The FHR pattern in the cardiotocographic recording is closely monitored for 1 to 10 minutes, using a 5-minute mean.
  Assess an acceleration of FHR defined as an increase in FHR ≥ 15 bpm (beats per minute for at least 15 seconds or normal FHR variability (5 to 25 bpm), or both. The presence of FHR acceleration or increased variability when previously reduced, or both, is interpreted as a positive response.
Differences in the results of intrapartum fetal scalp blood of fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in intrapartum pH results in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in newborn ph results of fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in newborn pH outcomes in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in the first minute apgar scores of the newborns in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in the minute-of-life Apgar scores of newborns in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in apgar scores at 5 minutes of life of newborns in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in apgar scores at 5 minutes of life of newborns in in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in the results of the type of newborn resuscitation in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in results of the type of newborn resuscitation in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in neonatal unit admission rates in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in the percentages of admission to the neonatal unit in fetuses with digital fetal scalp stimulations versus fetuses without digital fetal scalp stimulation
Differences in newborn seizure percentages in fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in newborn seizure percentages in fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation
Differences in the percentages of newborn deaths in fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation | 2 years
  Significant differences in percentages of newborn deaths in fetuses with digital fetal scalp stimulation vs. fetuses without digital fetal scalp stimulation
Differences in completion of cesarean delivery in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation. | 2 years
  Significant differences in completion of cesarean delivery in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation.
Differences in instrumental deliveries in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation. | 2 years
  Significant differences in instrumental deliveries in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation.
Differences in vaginal deliveries in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation. | 2 years
  Significant differences in vaginal deliveries in fetuses with digital fetal scalp stimulation versus fetuses without digital fetal scalp stimulation.
Percentage of fetuses with positive response to digital fetal scalp stimulation and intrapartum pH greater than 7.20 | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain an intrapartum pH greater than 7.20.
Percentage of fetuses with positive response to digital fetal scalp stimulation and intrapartum pH less than or equal to 7.20 | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain an intrapartum pH less than or equal to 7.20.
Percentage of fetuses with negative response to digital fetal scalp stimulation and intrapartum pH above 7.20. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain an intrapartum pH greater than 7.20.
Percentage of fetuses with negative response to digital fetal scalp stimulation and intrapartum pH less than or equal to 7.20. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain an intrapartum pH less than or equal to 7.20.
Percentage of fetuses with positive response to digital fetal scalp stimulation and neonatal pH above 7.20. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a neonatal pH greater than 7.20.
Percentage of fetuses with negative response to digital fetal scalp stimulation and neonatal pH above 7.20. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a neonatal pH greater than 7.20.
Percentage of fetuses with positive response to digital fetal scalp stimulation and neonatal pH less than or equal to 7.20. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a neonatal pH less than or equal to 7.20.
Percentage of fetuses with negative response to digital fetal scalp stimulation and neonatal pH less than or equal to 7.20. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a neonatal pH less than or equal to 7.20.
Percentage of fetuses with positive response to digital fetal scalp stimulation and apgar score greater than or equal to 8 in the first minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a apgar score greater than or equal to 8 in the first minute of life.
Percentage of fetuses with negative response to digital fetal scalp stimulation and apgar score greater than or equal to 8 in the first minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a apgar score greater than or equal to 8 in the first minute of life.
Percentage of fetuses with positive response to digital fetal scalp stimulation and apgar score less than 8 in the first minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a apgar score less than 8 in the first minute of life.
Percentage of fetuses with negative response to digital fetal scalp stimulation and apgar score less than 8 in the first minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a apgar score less than 8 in the first minute of life
Percentage of fetuses with a positive response to digital fetal scalp stimulation and an Apgar score greater than or equal to 8 at five minutes of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a apgar score greater than or equal to 8 at five minute of life
Percentage of fetuses with negative response to digital fetal scalp stimulation and apgar score greater than or equal to 8 at five minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a apgar score greater than or equal to 8 at five minute of life.Time Frame: 2 years
Percentage of fetuses with positive response to digital fetal scalp stimulation and apgar score less than 8 at five minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and obtain a apgar score less than 8 at five minute of life.
Percentage of fetuses with negative response to digital fetal scalp stimulation and apgar score less than 8 at five minute of life. | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and obtain a apgar score less than 8 at five minute of life
Percentage of fetuses with positive response to digital fetal scalp stimulation and type of neonatal resuscitation. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and the type of neonatal resuscitation.
Percentage of fetuses with negative response to digital fetal scalp stimulation and type of neonatal resuscitation. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and the type of neonatal resuscitation.
Percentage of fetuses with positive response to digital fetal scalp stimulation and requiring admission to the neonatal unit. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and require admission to the neonatal unit.
Percentage of fetuses with negative response to digital fetal scalp stimulation and requiring admission to the neonatal unit. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and require admission to the neonatal unit.
Percentage of fetuses with a positive response to digital fetal scalp stimulation who seizure | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being who respond positively to digital fetal scalp stimulation and who convulse.
Percentage of fetuses with a negative response to digital fetal scalp stimulation who seizure | 2 years
  To assess the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being who respond negatively to digital fetal scalp stimulation and who convulse.
Percentage of fetuses with positive response to digital fetal scalp stimulation and neonatal death. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond positively to digital fetal scalp stimulation and neonatal death.
Percentage of fetuses with negative response to digital fetal scalp stimulation and neonatal death. | 2 years
  To evaluate the percentage of fetuses with suspicious or pathologic cardiotocographic recording patterns compatible with risk of loss of fetal well-being that respond negatively to digital fetal scalp stimulation and neonatal death.

CONTACTS AND LOCATIONS:
Overall Officials: JAVIER PLAZA ARRANZ, Doctor, Study Director — Hospital Fundación Jiménez Diaz
Locations (2):
- Spain (2):
  - Fundación Jimenez Diaz Y Hospital La Zarzuela, Madrid
  - Hospital Universitario Sanitas La Zarzuela, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Practice Bulletin No. 106: Intrapartum fetal heart rate monitoring: nomenclature, interpretation, and general management principles. Obstet Gynecol. 2009 Jul;114(1):192-202. doi: 10.1097/AOG.0b013e3181aef106. No abstract available. PMID 19546798
- [Background] Murphy DJ, Shahabuddin Y, Yambasu S, O'Donoghue K, Devane D, Cotter A, Gaffney G, Burke LA, Molloy EJ, Boland F. Digital fetal scalp stimulation (dFSS) versus fetal blood sampling (FBS) to assess fetal wellbeing in labour-a multi-centre randomised controlled trial: Fetal Intrapartum Randomised Scalp Stimulation Trial (FIRSST NCT05306756). Trials. 2022 Oct 4;23(1):848. doi: 10.1186/s13063-022-06794-9. PMID 36195894
- [Background] Shakouri F, Iorizzo L, Edwards HMK, Vinter CA, Kristensen K, Isberg PE, Wiberg N. Effectiveness of fetal scalp stimulation test in assessing fetal wellbeing during labor, a retrospective cohort study. BMC Pregnancy Childbirth. 2020 Jun 5;20(1):347. doi: 10.1186/s12884-020-03030-7. PMID 32503518
- [Background] Tahmina S, Daniel M, Krishnan L. Manual fetal stimulation during intrapartum fetal surveillance: a randomized controlled trial. Am J Obstet Gynecol MFM. 2022 Mar;4(2):100574. doi: 10.1016/j.ajogmf.2022.100574. Epub 2022 Jan 17. PMID 35051669
- [Background] Al Wattar BH, Lakhiani A, Sacco A, Siddharth A, Bain A, Calvia A, Kamran A, Tiong B, Warwick B, MacMahon C, Marcus D, Long E, Coyle G, Lever GE, Michel G, Gopal G, Baig H, Price HL, Badri H, Stevenson H, Hoyte H, Malik H, Edwards J, Hartley J, Hemers J, Tamblyn J, Dalton JAW, Frost J, Subba K, Baxter K, Sivakumar K, Murphy K, Papadakis K, Bladon LR, Kasaven L, Manning L, Prior M, Ghosh M, Couch M, Altunel M, Pearce M, Cocker M, Stephanou M, Jie M, Mistry M, Wahby MO, Saidi NS, Ramshaw NL, Tempest N, Parker N, Tan PL, Johnson RL, Harris R, Tildesley R, Ram R, Painuly R, Cuffolo R, Bugeja R, Ngadze R, Grainger R, Gurung S, Mak S, Farrell S, Cowey S, Neary S, Quinn S, Nijjar SK, Kenyon S, Lamb S, Tracey S, Lee T, Kinsella T, Davidson T, Corr T, Sampson U, McQueen V, Smith WP, Castling Z; AB-FAB study group. Evaluating the value of intrapartum fetal scalp blood sampling to predict adverse neonatal outcomes: A UK multicentre observational study. Eur J Obstet Gynecol Reprod Biol. 2019 Sep;240:62-67. doi: 10.1016/j.ejogrb.2019.06.012. Epub 2019 Jun 15. PMID 31229725
- [Background] Carbonne B, Pons K, Maisonneuve E. Foetal scalp blood sampling during labour for pH and lactate measurements. Best Pract Res Clin Obstet Gynaecol. 2016 Jan;30:62-7. doi: 10.1016/j.bpobgyn.2015.05.006. Epub 2015 Jul 8. PMID 26253238
- [Background] Chandraharan E, Wiberg N. Fetal scalp blood sampling during labor: an appraisal of the physiological basis and scientific evidence. Acta Obstet Gynecol Scand. 2014 Jun;93(6):544-7. doi: 10.1111/aogs.12416. PMID 24806702
- [Background] Chandraharan E. Should national guidelines continue to recommend fetal scalp blood sampling during labor? J Matern Fetal Neonatal Med. 2016 Nov;29(22):3682-5. doi: 10.3109/14767058.2016.1140740. Epub 2016 Feb 24. PMID 26762827
- [Background] Tahir Mahmood U, O'Gorman C, Marchocki Z, O'Brien Y, Murphy DJ. Fetal scalp stimulation (FSS) versus fetal blood sampling (FBS) for women with abnormal fetal heart rate monitoring in labor: a prospective cohort study. J Matern Fetal Neonatal Med. 2018 Jul;31(13):1742-1747. doi: 10.1080/14767058.2017.1326900. Epub 2017 May 19. PMID 28475393
- [Background] Hughes O, Murphy DJ. Comparing second-line tests to assess fetal wellbeing in Labor: a feasibility study and pilot randomized controlled trial. J Matern Fetal Neonatal Med. 2022 Jan;35(1):91-99. doi: 10.1080/14767058.2020.1712704. Epub 2020 Jan 12. PMID 31928269
- [Background] East CE, Leader LR, Sheehan P, Henshall NE, Colditz PB, Lau R. Intrapartum fetal scalp lactate sampling for fetal assessment in the presence of a non-reassuring fetal heart rate trace. Cochrane Database Syst Rev. 2015 May 1;2015(5):CD006174. doi: 10.1002/14651858.CD006174.pub3. PMID 25929461
- [Background] Troha N, Razem K, Luzovec U, Lucovnik M. Comparison of Four Intrapartum Cardiotocography Classifications for Predicting Neonatal Acidemia at Birth. J Pregnancy. 2023 Feb 13;2023:5853889. doi: 10.1155/2023/5853889. eCollection 2023. PMID 36814692
- [Background] Alfirevic Z, Devane D, Gyte GM, Cuthbert A. Continuous cardiotocography (CTG) as a form of electronic fetal monitoring (EFM) for fetal assessment during labour. Cochrane Database Syst Rev. 2017 Feb 3;2(2):CD006066. doi: 10.1002/14651858.CD006066.pub3. PMID 28157275
- [Background] Murphy DJ, Devane D, Molloy E, Shahabuddin Y. Fetal scalp stimulation for assessing fetal well-being during labour. Cochrane Database Syst Rev. 2023 Jan 10;1(1):CD013808. doi: 10.1002/14651858.CD013808.pub2. PMID 36625680
- [Background] Jia YJ, Chen X, Cui HY, Whelehan V, Archer A, Chandraharan E. Physiological CTG interpretation: the significance of baseline fetal heart rate changes after the onset of decelerations and associated perinatal outcomes. J Matern Fetal Neonatal Med. 2021 Jul;34(14):2349-2354. doi: 10.1080/14767058.2019.1666819. Epub 2019 Sep 18. PMID 31533502
- See also: Fetal monitoring in labour — https://www.nice.org.uk/guidance/ng229
- See also: SEGO DOCUMENTOS DE CONSENSO 2007. — https://bibliotecavirtual.sego.es/protocolos